CLINICAL TRIAL: NCT04641754
Title: Phase II Clinical Study to Evaluate the Efficacy and Safety of WX-0593 in Patients With Crizotinib-resistant ALK -Positive, or Crizotinib-resistant/Crizotinib-naive ROS1-positive Non-small Cell Lung Cancer (NSCLC)
Brief Title: A Study Evaluates the Safety and Efficacy of WX-0593 in ALK -Positive, or ROS1-positive Non-small Cell Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WX0593-003
Record Dates: First submitted 2020-11-11; First posted 2020-11-24 (Actual); Last update posted 2020-11-24 (Actual); Status verified 2020-11

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- WX-0593 Tablets (Experimental): 60 mg of WX-0593 tablets, once daily for 7 days, followed by 180 mg of WX-0593 tablets, once daily in a 21-days cycle.
  Interventions: Drug: WX-0593 Tablets

INTERVENTIONS:
Drug: WX-0593 Tablets — tablets, 60 mg→180mg, quaque die（QD）
  Other Names: FL-006

SUMMARY:
The purpose of the study is to evaluate safety and efficacy of WX-0593 oral tablets in ALK -positive, or ROS1-positive non-small cell lung cancer (NSCLC)

DETAILED DESCRIPTION:
The clinical study is a single-arm, phase II, open label, multicenter design in patients with crizotinib-resistant ALK -positive, or crizotinib-resistant/crizotinib-naive ROS1-positive NSCLC.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years.
2. Female or male;
3. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2.
4. Expected survival no less than 12 weeks.
5. Patient should have at least one measurable lesion (RECIST 1.1); Lesions previously treated with radiotherapy can be considered target lesions only if there is a clear evidence of progression after radiotherapy.
6. Histologically or cytologically confirmed advanced ALK-positive NSCLC in upper first-class hospitals，or histologically or cytologically confirmed advanced ROS1-positive NSCLC in a central laboratory. Admission of ROS1-positive patients will be based on the positive test results confirmed by the central laboratory or by the local-approved method.

   1. Patients with ALK-positive NSCLC who had been progressive disease after at least 12 weeks of continuous treatment with crizotinib .
   2. Patients with ROS1-positive NSCLC who failed in standard treatment (eg.resistant /intolerance of crizotinib or chemotherapy).
   3. Patients with ROS1-positive NSCLC who cannot accept chemotherapy.
   4. ROS1-positive NSCLC patients who could not afford crizotinib treatment.
7. Patients with or without asymptomatic CNS metastases, or symptomatic brain metastasis after treatment stabilized for more than 4 weeks, and with stopping systemic sex hormone therapy for more than 2 weeks.
8. Organ functions should meet the following requirements (Blood components, cell growth factors, drugs that stimulate the growth of WBC or platelets, or drugs used to correct anemia are not permitted within 14 days prior to the laboratory examination): ANC≥1.5*10^9/L PLT≥90*10^9/L,Hb≥90 g/L, Total Bilirubin （TBIL）≤1.5*Upper Limit of Normal（ULN） ( Gilbert's Syndrome TBIL ≤3.0*ULN and DBIL≤1.5*ULN )，Alanine Transaminase （ALT）and Aspartate Aminotransferase （AST）≤2.5*ULN. For liver metastasis patients, ALT and AST≤5*ULN, Cr≤1.5*ULN, LVEF≥50%.
9. Any surgery, prior radiotherapy (except for palliative radiotherapy)/procedures must be completed at least 4 weeks prior to starting the treatment with study drug. Palliative radiotherapy must be completed within 48 hours prior to starting treatment.
10. Subject understands and voluntarily provides informed consent.

Exclusion Criteria:

1. Received any prior ALK inhibitors other than crizotinib.
2. Patients with brain meningeal metastasis.
3. Any clinically significant cardiovascular disease within 6 months prior to the first dose of the investigational drug, including but not limited to: myocardial infarction, severe/unstable angina, coronary artery/peripheral artery bypass graft, congestive heart failure, cerebrovascular accident (including transient ischemic attack).
4. Two consecutive corrected QT interval (QTc) > 480 ms through ECG examination during screening, patients with NCI-CTCAE v4.03 Grade ≥2 arrhythmia, Grade ≥2 heart failure, atrial fibrillation and ventricular fibrillation of any grade, or clinically significant supraventricular or ventricular arrhythmia requiring treatment or intervention.
5. Concomitant use of medications that may cause QTc prolongation or induce Torsades de pointes within 14 days prior to the first dose of the investigational drug or during treatment.
6. Continuous use of corticosteroids for more than 30 days, or require chronic use of corticosteroids or other immunosuppressants.
7. Past history of a large area of diffuse/interstitial pulmonary fibrosis, or known history of Grade 3 or 4 interstitial pulmonary fibrosis or interstitial lung disease, including a history of pneumonitis, hypersensitivity pneumonitis, interstitial pneumonitis, interstitial lung disease, obliterative bronchiolitis, or pulmonary fibrosis, but does not include local radiation pneumonitis or radiation-induced pulmonary fibrosis.
8. Patients with Grade > 1 nausea, vomiting, or diarrhea (CTCAE 4.03), other GI dysfunction or GI disease that may potentially affect drug absorption (such as ulcerative disease or malabsorption syndrome).
9. Subject received other clinical trial treatment within 1 month prior to the first dose of the investigational drug (if the medication received is a marketed drug, then refer to exclusion criteria #11).
10. Patients who are HBsAg-positive and/or HBcAb positive and HBV DNA >10^3 copies/mL, or HCV antibody-positive, or syphilis antibody- positive or known HIV infected.
11. No more than 2 weeks between the most recent use of another anti-cancer treatment (half life ≤3 days) and the first dose of the investigational drug, or the most recent use of another anti-cancer treatment (half life > 3 days) is less than 4 weeks. Patients previously treated with crizotinib could take WX-0593 tables after 1 week from the last dose.
12. Patients who cannot suspend the use of a strong CYP3A4 inducer or inhibitor at least 1 weeks prior to this study and during the study. These drugs include but are not limited to carbamazepine, phenobarbital, phenytoin, rifabutin, rifampicin, rifapentine, tipranavir, ritonavir, St. John's wart, and ketoconazole.
13. Patients who cannot suspend the use of a CYP3A4 substrate at least 1 weeks prior to this study and during the study, and the therapeutic index is low.
14. Pregnant or lactating female patients or a positive pregnancy test at baseline for females of childbearing potential.
15. Childbearing potential female patients who are unwilling to use effective contraceptive measures during the entire course of the study and within 6 months after the end of the study, or male patients who plan to have children.
16. Concurrent diseases that may seriously affect patient safety or impact patient completion of the study as determined by the investigator (such as clinically uncontrolled hypertension (blood pressure > 160/110 mmHg), severe diabetes, or thyroid disease).
17. Drug or alcohol abuse. Alcohol abuse refers to drinking 14 units of alcohol per week: 1 unit = 285mL of beer, or 25mL of spirits, or 100mL of wine.
18. History of definitive neurological or mental disorder, including epilepsy or dementia.
19. Patients with other malignant tumors within 3 years prior to screening (except for cured basal cell carcinoma of the skin, cervical carcinoma in situ, thyroid carcinoma in situ, and papillary thyroid carcinoma).
20. Patients with added risks associated with the study or may interfere with the interpretation of study results as determined by the investigator, or deemed unsuitable by the investigator and/or sponsor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Estimated)
Dates: Start 2019-03-07 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Confirmed Objective Response Rate (ORR) Assessed By An Independent Review Committee | From frist administration of WX-0593 to the date that the last patients observed for 18 weeks.
  ORR is defined the percentage of the participants who are confirmed to have achieved complete response (CR) or partial response (PR) per an Independent Review Committee (IRC) using Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 after the initiation of study treatment.

SECONDARY OUTCOMES:
Confirmed Objective Response Rate (ORR) Assessed By Investigators | From frist administration of WX-0593 to the date that the last patients observed for 18 weeks.
  ORR is defined the percentage of the participants who are confirmed to have achieved complete response (CR) or partial response (PR) per Investigators using Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 after the initiation of study treatment.
Progression-free survival (PFS) | From frist administration of WX-0593 until firstly recorded disease progression or death (whichever occurs earlier), or to the date that the last patients observed for 18 weeks.
  PFS defined as the time from baseline to first observed disease progression or death from any cause.
Disease Control Rate (DCR) | From frist administration of WX-0593 to the date that the last patients observed for 18 weeks.
  DCR is the percentage of patients with best response of CR, PR or Stable Disease (SD).
Duration of Response (DOR) | From frist administration of WX-0593 to the date that the last patients observed for 18 weeks .
  The DOR is defined as the time from the date of the first response CR/PR (whichever is first recorded) to the date on which progressive disease (PD) is first noted or date of death.
Time to Progression (TTP) | From frist administration of WX-0593 to the date that the last patients observed for 18 weeks.
  Time to Progression
Confirmed Intracranial Objective Response Rate (iORR) | From frist administration of WX-0593 to the date that the last patients observed for 18 weeks.
  Confirmed iORR is defined as the proportion of the participants who have achieved CR or PR in the brain per a modification of RECIST version 1.1, after the initiation of study treatment, in participants with intracranial brain metastases at baseline.
Overall Survival (OS) | From frist administration of WX-0593 until death due to any cause, withdraws informed consent, is lost to follow-up or refuses phone visits, or study completion（up to 2.5 years）
  OS is the time from the start of study treatment to the date of death.
Incidence of Adverse Events | the date of written informed consent signed until at least 28 days after the last dose of study drug was administered.
  Incidence of All Adverse Events, Serious Adverse Events and Treatment-Emergent Adverse Events by CTCAE v4.03
Cssmin | Pre-dose on Cycle 1 Day 1, Cycle 1 Day 7, Cycle 1 Day 21, Cycle 2 Day 21, and Cycle 4 Day 21 (each cycle is 21 days)
  Minimum value of steady plasma-drug concentration for WX-0593

CONTACTS AND LOCATIONS:
Locations (41):
- China (41):
  - The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - Oncology Department, Anhui Cancer Hospital, Hefei, Anhui
  - Respiratory Department, Anhui Cancer Hospital, Hefei, Anhui
  - Cancer Institute and Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Chinese PLA General Hospital, Beijing, Beijing Municipality
  - Thoracic Oncology I Department, Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Thoracic Oncology II Department, Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Beijing Chest Hospital, Beijing, Beijing Municipality
  - General Department, Beijing Chest Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Army Medical Center of PLA, Chongqing, Chongqing Municipality
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Gansu Cancer Hospital, Lanzhou, Gansu
  - Cancer Center of Guangzhou Medical University, Guangzhou, Guangdong
  - Liuzhou People's Hospital, Liuchow, Guangxi
  - The Fourth Hospital of Hebei Medical University, Shijiangzhuang, Hebei
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Hunan Tumor Hospital, Changsha, Hunan
  - The Affiliated Hospital of Inner Mongolia Medical University, Hohhot, Inner Mongolia
  - Nanjing Chest Hospital, Nanjing, Jiangsu
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - The Affiliated Hospital of Jiangnan University, Wuxi, Jiangsu
  - Xuzhou Central Hospital, Xuzhou, Jiangsu
  - The First Hospital of Jilin University, Changchun, Jilin
  - Jilin Cancer Hospital, Changchun, Jilin
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Jinan Central Hospital, Jinan, Shandong
  - Shandong Cancer Hospital, Jinan, Shandong
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - Yantai Yuhuangding Hospital, Yantai, Shandong
  - Shanxi Cancer Hospital, Taiyuan, Shanxi
  - Tangdu Hospital, Xi’an, Shanxi
  - Affiliated Hospital of North Sichuan Medical College, Nanchong, Sichuan
  - Tianjin Cancer Hospital, Tianjin, Tianjin Municipality
  - Cancer Hospital Affiliated to Xinjiang Medical University, Ürümqi, Xinjiang
  - Yunnan Cancer Hospital, Kunming, Yunnan
  - Hangzhou first people's Hospital, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang

REFERENCES:
- [Derived] Shi Y, Chen J, Zhang H, Zhang Z, Zhang Y, Wang Z, Zhang S, Zhao J, Liu C, Wang X, Zhao Y, Hu C, Yang L, Hao X, Wang L, Liu Y, Yu Y, Zhao J, Wang M, Zhang L, Sun S, Hu Y, Gu K, Hang X, Shan J, Zhang Y, Tan B, Yang W, Yang R, Si M, Geng H, Li H, Kang X. Efficacy and safety of iruplinalkib (WX-0593) in ALK-positive crizotinib-resistant advanced non-small cell lung cancer patients: a single-arm, multicenter phase II study (INTELLECT). BMC Med. 2023 Feb 24;21(1):72. doi: 10.1186/s12916-023-02738-5. PMID 36829154